CLINICAL TRIAL: NCT02300025
Title: A Study to Evaluate the Pharmacokinetics and Safety of Cobimetinib in Volunteers With and Without Liver Damage
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: GP29342
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-01

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — cobimetinib

ARMS (4):
- Cohort 1: Normal function (Experimental)
  Interventions: Drug: cobimetinib
- Cohort 2: Mild Hepatic Impairment (Experimental)
  Interventions: Drug: cobimetinib
- Cohort 3: Moderate Hepatic Impairment (Experimental)
  Interventions: Drug: cobimetinib
- Cohort 4: Severe Hepatic Impairment (Experimental)
  Interventions: Drug: cobimetinib

INTERVENTIONS:
Drug: cobimetinib — single oral 10-mg dose of cobimetinib

SUMMARY:
This study is an open-label, multi-center, single-dose, parallel group study to determine the pharmacokinetics, safety, and tolerability of cobimetinib administered at 10 mg to fasted male and female adult subjects with varying degrees of hepatic function. The study will be conducted based on the Child-Pugh classification of hepatic impairment. The anticipated duration of the study is 7.5 weeks. The target sample sizes are: 18 volunteers with varying degrees of hepatic function and up to 12 healthy control volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 74 years of age, inclusive
* Body weight >/=45 kg and body mass index between 17 and 41 kg/m2, inclusive
* Subjects with hepatic impairment must have a Child-Pugh score of 5 to 6 (mild), 7 to 9 (moderate), or 10 to 15 (severe) and have stable hepatic insufficiency within 1 month prior to Screening and a stable medication regimen for at least 1 month prior to Check-in
* Agreement to use highly effective contraceptive methods as defined in the protocol

Exclusion Criteria:

* Significant illness, including infections, or hospitalization within the 2 weeks prior to dosing, except for subjects with hepatic impairment who due to their liver disease may be affected by significant medical problems which require frequent hospitalizations. Invasive systemic fungal infections need to be fully treated prior to study entry
* Significant history or clinical manifestations of any cardiac event that would put the subject at risk in the opinion of the Investigator
* Use of drugs of abuse within 1 month of Screening or during the entire study
* Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United States (3):
  - Anaheim, California
  - Miami, Florida
  - Orlando, Florida

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Normal Hepatic Function: Participants with normal hepatic function received single oral dose of 10 milligrams (mg) cobimetinib (two 5 mg capsules) on Day 1 of study.
- Cohort 2: Mild Hepatic Impairment: Participants with mild hepatic impairment (Child-Pugh Class A, score of 5 to 6, inclusive) received single oral dose of 10 mg cobimetinib (two 5 mg capsules) on Day 1 of study.
- Cohort 3: Moderate Hepatic Impairment: Participants with moderate hepatic impairment (Child-Pugh Class B, score of 7 to 9, inclusive) received single oral dose of 10 mg cobimetinib (two 5 mg capsules) on Day 1 of study.
- Cohort 4: Severe Hepatic Impairment: Participants with severe hepatic impairment (Child-Pugh Class C, score of 10 to 15, inclusive) received single oral dose of 10 mg cobimetinib (two 5 mg capsules) on Day 1 of study.
Period: Overall Study
Arm/Group | Cohort 1: Normal Hepatic Function | Cohort 2: Mild Hepatic Impairment | Cohort 3: Moderate Hepatic Impairment | Cohort 4: Severe Hepatic Impairment
Started | 10 | 6 | 6 | 6
Completed | 10 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of cobimetinib and had at least one post-dose safety assessment.
Groups:
- Cohort 1: Normal Hepatic Function: Participants with normal hepatic function received single oral dose of 10 mg cobimetinib (two 5 mg capsules) on Day 1 of study.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Normal Hepatic Function | Cohort 2: Mild Hepatic Impairment | Cohort 3: Moderate Hepatic Impairment | Cohort 4: Severe Hepatic Impairment | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56 (6.8) | 59 (2.8) | 61 (2.9) | 53 (5.3) | 57 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 2 | 9
  Male | 7 | 3 | 5 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Pre-dose (0 hours [hrs]), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 264, 336, 456, and 576 hrs post-dose
Population: Pharmacokinetic (PK) population included all participants who received at least one dose of cobimetinib and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Cohort 1: Normal Hepatic Function | Cohort 2: Mild Hepatic Impairment | Cohort 3: Moderate Hepatic Impairment | Cohort 4: Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 6 | 6 | 6
nanograms per milliliter (ng/mL) | 10.7 (7.41) | 9.00 (4.09) | 8.03 (2.49) | 3.97 (1.77)
Statistical Analysis 1: Comparison: Cohort 1: Normal Hepatic Function vs Cohort 2: Mild Hepatic Impairment; Cmax was analyzed using a mixed model analysis of variance (ANOVA) to determine 90% confidence interval (CI) of the ratio between normal hepatic function (reference) and mild hepatic impairment (test) where hepatic impairment group was a fixed factor. The least squares (LS) means of the test and reference treatments obtained from the mixed model were back-transformed to give geometric LS means (a point estimate); Test type: Superiority or Other; LS means ratio = 92.2, 90% CI 2-sided [59.2 to 143.4] — The 90% CI for differences in LS means between test and reference treatments obtained from mixed model were also back-transformed to give 90% CIs for the ratio of the test treatment relative to the reference treatment
Statistical Analysis 2: Comparison: Cohort 1: Normal Hepatic Function vs Cohort 3: Moderate Hepatic Impairment; Cmax was analyzed using a mixed model ANOVA to determine 90% CI of the ratio between normal hepatic function (reference) and moderate hepatic impairment (test) where hepatic impairment group was a fixed factor. The LS means of the test and reference treatments obtained from the mixed model were back-transformed to give geometric LS means (a point estimate); Test type: Superiority or Other; LS means ratio = 84.9, 90% CI 2-sided [54.6 to 132.1] — The 90% CI for differences in LS means between the test and reference treatments obtained from the mixed model were also back-transformed to give 90% CIs for the ratio of the test treatment relative to the reference treatment
Statistical Analysis 3: Comparison: Cohort 1: Normal Hepatic Function vs Cohort 4: Severe Hepatic Impairment; Cmax was analyzed using a mixed model ANOVA to determine 90% CI of the ratio between normal hepatic function (reference) and severe hepatic impairment (test) where hepatic impairment group was a fixed factor. The LS means of the test and reference treatments obtained from the mixed model were back-transformed to give geometric LS means (a point estimate); Test type: Superiority or Other; LS means ratio = 39.0, 90% CI 2-sided [25.1 to 60.7] — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: Pre-dose (0 hrs), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 264, 336, 456, and 576 hrs post-dose
Population: PK population.
Measure: Median (Full Range); unit: hrs
Arm/Group | Cohort 1: Normal Hepatic Function | Cohort 2: Mild Hepatic Impairment | Cohort 3: Moderate Hepatic Impairment | Cohort 4: Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 6 | 6 | 6
hrs | 2 [1 to 6] | 6 [2 to 6] | 4 [2 to 6] | 2 [1 to 4]

3. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)]
Description: AUC (0-t) was defined as area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t).
Time Frame: Pre-dose (0 hrs), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 264, 336, 456, and 576 hrs post-dose
Population: PK Population.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1: Normal Hepatic Function | Cohort 2: Mild Hepatic Impairment | Cohort 3: Moderate Hepatic Impairment | Cohort 4: Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 6 | 6 | 6
ng*hr/mL | 604 (606) | 498 (200) | 539 (296) | 268 (181)
Statistical Analysis 1: Comparison: Cohort 1: Normal Hepatic Function vs Cohort 2: Mild Hepatic Impairment; AUC (0-t) was analyzed using a mixed model ANOVA to determine 90% CI of the ratio between normal hepatic function (reference) and mild hepatic impairment (test) where, hepatic impairment group was a fixed factor. The LS means of the test and reference treatments obtained from the mixed model were back-transformed to give geometric LS means (a point estimate); Test type: Superiority or Other; LS means ratio = 98.4, 90% CI 2-sided [52.0 to 186.0] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Cohort 1: Normal Hepatic Function vs Cohort 3: Moderate Hepatic Impairment; AUC (0-t) was analyzed using a mixed model ANOVA to determine 90% CI of the ratio between normal hepatic function (reference) and moderate hepatic impairment (test) where, hepatic impairment group was a fixed factor. The LS means of the test and reference treatments obtained from the mixed model were back-transformed to give geometric LS means (a point estimate); Test type: Superiority or Other; LS means ratio = 102.2, 90% CI 2-sided [54.0 to 193.2] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Cohort 1: Normal Hepatic Function vs Cohort 4: Severe Hepatic Impairment; AUC (0-t) was analyzed using a mixed model ANOVA to determine 90% CI of the ratio between normal hepatic function (reference) and severe hepatic impairment (test) where, hepatic impairment group was a fixed factor. The LS means of the test and reference treatments obtained from the mixed model were back-transformed to give geometric LS means (a point estimate); Test type: Superiority or Other; LS means ratio = 42.5, 90% CI 2-sided [22.5 to 80.5] — [estimate comment as in outcome 1, analysis 2]

4. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]
Description: AUC (0 - ∞) was defined as AUC from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t- ∞).
Time Frame: Pre-dose (0 hrs), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 264, 336, 456, and 576 hrs post-dose
Population: PK population. Here, number of participants analyzed signified those participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1: Normal Hepatic Function | Cohort 2: Mild Hepatic Impairment | Cohort 3: Moderate Hepatic Impairment | Cohort 4: Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 6 | 6 | 5
ng*hr/mL | 637 (606) | 530 (206) | 579 (301) | 370 (163)
Statistical Analysis 1: Comparison: Cohort 1: Normal Hepatic Function vs Cohort 2: Mild Hepatic Impairment; AUC (0 - ∞) was analyzed using a mixed model ANOVA to determine 90% CI of the ratio between normal hepatic function (reference) and mild hepatic impairment (test) where hepatic impairment group was a fixed factor. The LS means of the test and reference treatments obtained from the mixed model were back-transformed to give geometric LS means (a point estimate); Test type: Superiority or Other; LS means ratio = 97.6, 90% CI 2-sided [59.3 to 160.6] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Cohort 1: Normal Hepatic Function vs Cohort 3: Moderate Hepatic Impairment; AUC (0 - ∞) was analyzed using a mixed model ANOVA to determine 90% CI of the ratio between normal hepatic function (reference) and moderate hepatic impairment (test) where hepatic impairment group was a fixed factor. The LS means of the test and reference treatments obtained from the mixed model were back-transformed to give geometric LS means (a point estimate); Test type: Superiority or Other; LS means ratio = 103.0, 90% CI 2-sided [62.6 to 169.6] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Cohort 1: Normal Hepatic Function vs Cohort 4: Severe Hepatic Impairment; AUC (0 - ∞) was analyzed using a mixed model ANOVA to determine 90% CI of the ratio between normal hepatic function (reference) and severe hepatic impairment (test) where hepatic impairment group was a fixed factor. The LS means of the test and reference treatments obtained from the mixed model were back-transformed to give geometric LS means (a point estimate); Test type: Superiority or Other; LS means ratio = 68.5, 90% CI 2-sided [40.4 to 116.2] — [estimate comment as in outcome 1, analysis 2]

5. Primary Outcome: Extrapolated Area Under the Curve (AUC Percent [%] Extrapolated)
Description: AUC% extrapolated was defined as the percentage of AUC [0-∞] obtained by forward extrapolation. It is calculated as [AUC (0-∞) minus AUC(0-t]*100/ AUC (0-∞), where AUC [0-∞] = Area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (0-∞) and AUC(0-t) is area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration.
Time Frame: Pre-dose (0 hrs), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 264, 336, 456, and 576 hrs post-dose
Population: PK population. Here, number of participants analyzed signified those participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: % extrapolated
Arm/Group | Cohort 1: Normal Hepatic Function | Cohort 2: Mild Hepatic Impairment | Cohort 3: Moderate Hepatic Impairment | Cohort 4: Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 6 | 6 | 5
% extrapolated | 7.37 (4.37) | 6.69 (2.63) | 8.17 (4.36) | 15.90 (4.79)

6. Primary Outcome: Apparent Terminal Elimination Rate Constant (λZ)
Description: λZ was defined as the magnitude of the slope of the linear regression of the log concentration versus time profile during the terminal phase.
Time Frame: Pre-dose (0 hrs), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 264, 336, 456, and 576 hrs post-dose
Population: PK population. Here, number of participants analyzed signified those participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: 1 per hr (1/hr)
Arm/Group | Cohort 1: Normal Hepatic Function | Cohort 2: Mild Hepatic Impairment | Cohort 3: Moderate Hepatic Impairment | Cohort 4: Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 6 | 6 | 5
1 per hr (1/hr) | 0.00942 (0.00259) | 0.00852 (0.00315) | 0.00702 (0.00181) | 0.00509 (0.00114)

7. Primary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration of cobimetinib to decrease by one half.
Time Frame: Pre-dose (0 hrs), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 264, 336, 456, and 576 hrs post-dose
Population: PK population. Here, number of participants analyzed signified those participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Cohort 1: Normal Hepatic Function | Cohort 2: Mild Hepatic Impairment | Cohort 3: Moderate Hepatic Impairment | Cohort 4: Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 6 | 6 | 5
hr | 79.1 (22.7) | 95.2 (48.2) | 104.0 (24.4) | 143.0 (40.4)

8. Primary Outcome: Apparent Oral Clearance (CL/F)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Pre-dose (0 hrs), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 264, 336, 456, and 576 hrs post-dose
Population: PK population. Here, number of participants analyzed signified those participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: Liter per hr (L/hr)
Groups:
- Cohort 4: Severe Hepatic Impairment: Participants with severe hepatic impairment received single oral dose of 10 mg cobimetinib (two 5 mg capsules) on Day 1 of study.
Arm/Group | Cohort 1: Normal Hepatic Function | Cohort 2: Mild Hepatic Impairment | Cohort 3: Moderate Hepatic Impairment | Cohort 4: Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 6 | 6 | 5
Liter per hr (L/hr) | 23.4 (11.6) | 22.9 (13.2) | 21.9 (11.7) | 31.7 (14.5)

9. Primary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/F after the oral dose is influenced by the fraction absorbed.
Time Frame: Pre-dose (0 hrs), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, 216, 264, 336, 456, and 576 hrs post-dose
Population: PK population. Here, number of participants analyzed signified those participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Cohort 1: Normal Hepatic Function | Cohort 2: Mild Hepatic Impairment | Cohort 3: Moderate Hepatic Impairment | Cohort 4: Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 6 | 6 | 5
Liter | 2580 (1300) | 2880 (1370) | 3230 (1650) | 6280 (2480)

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of study drug (up to approximately 2 months)
Groups:
- Cohort 4: Severe Hepatic Impairment: Participants with severe hepatic impairment (Child-Pugh Class A, score of 10 to 15, inclusive) received single oral dose of 10 mg cobimetinib (two 5 mg capsules) on Day 1 of study.
Arm/Group | Cohort 1: Normal Hepatic Function | Cohort 2: Mild Hepatic Impairment | Cohort 3: Moderate Hepatic Impairment | Cohort 4: Severe Hepatic Impairment
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/10 | 3/6 | 2/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Normal Hepatic Function (N=10) | Cohort 2: Mild Hepatic Impairment (N=6) | Cohort 3: Moderate Hepatic Impairment (N=6) | Cohort 4: Severe Hepatic Impairment (N=6)
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.